CLINICAL TRIAL: NCT06584409
Title: The Comparsion of Primary Headache in Blood Test of MMP2 and CGRP: A Single Blind Randomized Sham-laser-acupuncture Controlled Study.
Brief Title: Migraines Accepted Laser Acupuncture Compared in Blood Test of MMP2 and CGRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CF24162B
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-08

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Observation

STUDY DESIGN:
Intervention Model Description: The patients was divided to sham group or laser acupuncture group. After 1 months treatment, and followed up for 6 months., the sham group received complementary laser acupuncture for 1 months and followed up for another 3 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were randomized by computer software (Excel 2016 for Windows) and the randomization process was overseen by the Institutional Review Board at Taichung Veterans General Hospital. All the participants and our collaborative case-manager were blinded to treatment types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Experimental): CM patients with unsatisfactory pharmacological effects receive laser acupuncture for 8 sessions that spanned 4 weeks. Laser stimulation energy of 4.5 J for 30 seconds at each of the following acupoints: bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3)
  Interventions: Device: Laser Pen
- Sham treatment (Sham Comparator): CM patients with unsatisfactory pharmacological effects receive sham treatment for 8 sessions that spanned 4 weeks. Sham treatment had no laser output.
  Interventions: Other: Observation

INTERVENTIONS:
Device: Laser Pen — Laser stimulation energy of 4.5 J for 30 seconds at each of the following acupoints: bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3)
  Arms: Laser treatment
Other: Observation — Sham treatment with no laser output, stimulate the same acupoints as laser acupuncture group as follows: 30 seconds at bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3)
  After 6 months followed up, the sham group received truely Laser stimulation energy of 4.5 J for 30 seconds at each of the following acupoints: bilateral Cuanzhu (BL2), Fengchi (GB20), Taiyang (EX-HN5), Shuaigu (GB8), Hegu (LI4), Taichong (LR3) and midline Yintang (EX-HN3), and followed up for another 3 months.
  Arms: Sham treatment

SUMMARY:
Aims:

To investigate the efficacy of laser-acupuncture for the severity of primary headache and comorbidities, and the Lab data examination.

Methods:

In this hospital-based prospective single blind randomized sham-controlled study, patients over 18 years old with primary headache will be randomly divided into two treatment arms including laser-acupuncture and sham-controlled group. The expected laser-acupuncture protocol will be bilateral BL2, GB20, EX-HN5, GB8, LI4, LR3 and midline EX-HN3 in totally eight sessions at the first month. In the sham-laser-acupuncture group, patients will receive eight sessions of laser-acupuncture for free after unblinding. We expected to track patients for at least half year. The diagnosis and classification of headache was evaluated using the ICHD-3 criteria. The severity of headache was evaluated using Migraine Disability Assessment (MIDAS) and headache diary provided by Taiwan Headache Society. The co-primary efficacy end points are change in migraine days per month and variation of MIDAS. The secondary end point is the reducing of the severity of comorbidities including headache related anxiety and depression, and both of the quality of life and sleep.

In addition, patients' characteristics will be investigated as follows:

1. Sociodemographic factors (ethnicity, age, sex, body weight, BMI, blood pressure)
2. Headache related parameters (onset, duration, pain scale, current medication for headache, menstrual cycle)
3. Anxiety, evaluate by Hospital Anxiety and Depression Scale (HADS)
4. Depression, evaluate by Beck's Depression Inventory
5. Quality of life, evaluate by 36-Item Short Form Survey (SF-36)
6. Quality of sleep, evaluate by Pittsburgh Sleep Quality Index (PSQI)
7. Aura of headache
8. Episodic or chronic headache (If patient diagnosed as migraine.)
9. Nausea, vomiting, photophobia, phonophobia (If patient diagnosed as migraine.) During the following time, we will need the patient's blood samples four times, each times 20cc, all need 80cc for Lab test of MMP2, CGRP, substance P, beta-endorphin.

Importance:

In our hospital, we perform laser-acupuncture for patients with headache for several years. A prospective randomized controlled study is the key tools to establish the efficacy of laser-acupuncture for primary headache, and the Lab data with MMP2, CGRP, substance P, beta-endorphin for approval. Look forward to help improve therapeutic strategies in clinical practice.

DETAILED DESCRIPTION:
Headache is one of the most common complaints encountered in medical institution as known as an almost universal human experience. Approximately 65% of headaches are classified as primary, which was a composite of migraine, tension-type headache, trigeminal autonomic cephalalgia and other primary headaches according to the third edition of the International Classification of Headache Disorders (ICHD-3). Primary headaches encompass a heterogeneous group of neurologic disorders and might be bothersome for patients.

It's well established that acupuncture can be considered a treatment option for migraine prevention. The efficacy of laser-acupuncture is similar to acupuncture, and laser-acupuncture is a non-invasive therapeutic approach and safety. It could reduce the risk of hemorrhage, infection and needle phobia. However, the efficacy of laser-acupuncture in primary headache remains inconclusive.

MMP2, CGRP, substance P, beta-endorphin are new Lab examination for following up the patients suffered from migraine.

Aims:

To investigate the efficacy of laser-acupuncture for the severity of primary headache and comorbidities, and the Lab data examination.

Methods:

In this hospital-based prospective single blind randomized sham-controlled study, patients over 18 years old with primary headache will be randomly divided into two treatment arms including laser-acupuncture and sham-controlled group. The expected laser-acupuncture protocol will be bilateral BL2, GB20, EX-HN5, GB8, LI4, LR3 and midline EX-HN3 in totally eight sessions at the first month. In the sham-laser-acupuncture group, patients will receive eight sessions of laser-acupuncture for free after unblinding. We expected to track patients for at least half year. The diagnosis and classification of headache was evaluated using the ICHD-3 criteria. The severity of headache was evaluated using Migraine Disability Assessment (MIDAS) and headache diary provided by Taiwan Headache Society. The co-primary efficacy end points are change in migraine days per month and variation of MIDAS. The secondary end point is the reducing of the severity of comorbidities including headache related anxiety and depression, and both of the quality of life and sleep.

In addition, patients' characteristics will be investigated as follows:

1. Sociodemographic factors (ethnicity, age, sex, body weight, BMI, blood pressure)
2. Headache related parameters (onset, duration, pain scale, current medication for headache, menstrual cycle)
3. Anxiety, evaluate by Hospital Anxiety and Depression Scale (HADS)
4. Depression, evaluate by Beck's Depression Inventory
5. Quality of life, evaluate by 36-Item Short Form Survey (SF-36)
6. Quality of sleep, evaluate by Pittsburgh Sleep Quality Index (PSQI)
7. Aura of headache
8. Episodic or chronic headache (If patient diagnosed as migraine.)
9. Nausea, vomiting, photophobia, phonophobia (If patient diagnosed as migraine.) During the following time, we will need the patient's blood samples four times, each times 20cc, all need 80cc for Lab test of MMP2, CGRP, substance P, beta-endorphin.

Importance:

In our hospital, we perform laser-acupuncture for patients with headache for several years. A prospective randomized controlled study is the key tools to establish the efficacy of laser-acupuncture for primary headache, and the Lab data with MMP2, CGRP, substance P, beta-endorphin for approval. Look forward to help improve therapeutic strategies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patient under the diagnosis and classification of headache was evaluated using the ICHD-3 criteria.

Exclusion Criteria:

* Age under 18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
cGRP | 12 weeks, 24 weeks, 36 weeks
  change in cGRP from baasline and each follow-up time point
MMP2 | 12 weeks, 24 weeks, 36 weeks
  change in MMP2 from baasline and each follow-up time point

SECONDARY OUTCOMES:
Difference in the number of headache days per month | 12 weeks, 24 weeks, 36 weeks
  change in monthly migraine days (MMD) from baseline and each follow-up time point
Difference in the of headache attacks lasting hours per month | 12 weeks, 24 weeks, 36 weeks
  change in acute headache medications usage days per month from baseline and each follow-up time point
Difference in the headache pain intensity (NRS) | 12 weeks, 24 weeks, 36 weeks
  changes in the headache severity (based on NRS) between baseline and each follow-up time point
Difference in the number of days with acute headache medication intake per month | 12 weeks, 24 weeks, 36 weeks
  change in acute headache medications usage days per month from baseline and each follow-up time point
Difference in the Migraine Disability Assessment | 12 weeks, 24 weeks, 36 weeks
  changes in the Migraine Disability Assessmen between baseline and each follow-up time point.
  Title: Migraine Disability Assessmen Maximum value:450 Minimum value:0 Higher scores mean: worsen outcome
Difference in the Beck's Depression Inventory | 12 weeks, 24 weeks, 36 weeks
  change in Beck's Depression Inventory between baseline and each follow-up time point
  Title:Beck's Depression Inventory Maximum value:63 Minimum value:0 Higher scores mean: worsen outcome
Difference in the Hospital Anxiety and Depression Scale | 12 weeks, 24 weeks, 36 weeks
  change in Hospital Anxiety and Depression Scale between baseline and each follow-up time point
  Title:Hospital Anxiety and Depression Scale Maximum value:21/21 Minimum value:0/0 Higher scores mean:worsen outcome
30% reduction in migraine days | 12 weeks, 24 weeks, 36 weeks
  ≥ 30% reduction in migraine days between baseline and each follow-up time point
Substance P | 12 weeks, 24 weeks, 36 weeks
  change in Substance P from baasline and each follow-up time point
beta-endorphin | 12 weeks, 24 weeks, 36 weeks
  change in beta-endorphin from baasline and each follow-up time point

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hsiang Chou, M.D., Principal Investigator — Taichung Veterans General Hospital; Chi Sheng Wang, M.D., Study Director — Taichung Veterans General Hospital; Huan Yun Wu, M.D., Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichang, Taiwan

IPD SHARING:
Plan to Share IPD: No